CLINICAL TRIAL: NCT03118128
Title: Effect of the Addition of Metformin Hydrochloride on the Prognosis of Patients With B-cell Precursor (Ph+ Negative) Acute Lymphoblastic Leukemia With High Expression of ABCB1 Gene
Brief Title: Metformin Reduce the Relapse Rate on Patients With B-cell Precursor (Ph+ Negative) Acute Lymphoblastic Leukemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital General de Mexico (Other Government)
Responsible Party: Principal Investigator, Christian Ramos Penafiel, Principal Investigator, Hospital General de Mexico
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HGM-CRP2-LLA
Record Dates: First submitted 2017-04-07; First posted 2017-04-18 (Actual); Last update posted 2017-07-06 (Actual); Status verified 2017-04

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Acute Lymphoblastic Leukemia (ALL), ABCB1, Metformin
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- metformin (Active Comparator): Metformin 850mg PO three times a day, during the pre-induction with steroids, induction remission, consolidation and maintenance
  Interventions: Drug: Metformin
- No metformin (No Intervention)

INTERVENTIONS:
Drug: Metformin — Metformin 850 mg PO three times a day plus prednisone in one 7-days cycle as pre-treatment and during the 28 days induction remission treatment, consolidation therapy and maintenance
  Arms: metformin

SUMMARY:
Metformin's Antitumor activity were identified from differens diabetic patients trials, mainly associated to its mechanism of action and protein - kinase AMPK (AMP-activated protein kinase) activation. According to Cancer and Diabetes International Consensus from 2012, diabetes increases the risk for developping cancer and metformin has an protector effect against cancer cells and has an impact on overall survival.

Chemotherapy drug resistance induces treatment fail in oncology. Metformin increases AMPK levels, blocks PI3K (phosphatidylinositol 3- kinase)/ AKT /mTOR(mammailian Target of Rapamycin) pathway but few evidence associated with drug resistance gene expression.

This is an, experimental one-center study that pretends to stablish the effect of adding metformin 850 mg PO three times a day over the multi-drug resistance gene expression (ABCB1) in de novo Acute Lymphoblastic Leukemia in one 7-days cycle with prednisone as pre-treatment- and on the induction remission treatment.

DETAILED DESCRIPTION:
The MDR (Multidrug-Resistance) Genes are implicated on the resistance of several types of cancer. The most important on leukemia are the ABCB1 and ABCG2- ABCB1 are implicated on resistance and severity on Acute Myeloid Leukemia and pediatric Acute Lymphoblastic Leukemia. Those transporters use ATP for use. Metformin decrease the intracellular ATP (Adenosine triphosphate) reserve the by the activation of AMPK. Recently on MCF7-Adr (Michigan Cancer Foundation 7, breast cancer cell line) cancer cell line, Metformin block the function of the P-glycoprotein by the inhibition of the Nuclear Factor -kappa-B.

The clinical evidence at this moment is limited, based on small clinical trials or observational studies. This study tries to evaluate the effect of the addition of Metformin to a standard chemotherapy regimen on patients who express high levels of expression of mRNA (messenger ribonucleic acid) ABCB1

Experimental protocol

The patients will be stratified on three groups: The high-expression, low expression and absent gene expression according the level mRNA of ABCB1 at diagnostic. The samples are obtained from mononuclear peripheral blood cells

Extraction of total RNA Total RNA was isolated by TRIzol® (Invtirogen Life Technologies) according to the manufacturer´s recomendations described by Chomczynski and Sacchi.

The concentration and purity of total RNA was determined in a UV -vis spectrophotometer (Thermo Scientific , Genesis 10S UV-vis). The integrity of the genetic material was confirmed by 1.5% agarose gel electrophoresis at 70 V for 40 min. The RNA was stored at -80°C until needed.

Synthesis of cDNA Fort he synthesis of c DNA (complementary deoxyribonucleic acid) the amount of RNA used was 2µg for a final volume of 20 µg. The RNA was mixed with 1 µl oligonucleotide 12-18 (INVITROGEN, Carlsbad, CA) and 1 µl de dNTPs (deoxynucleoside triphosphate) 10mM (Applied Biosystems, Roche). After the addition of 4 µl of Buffer 5 X (Tris- HCl (hydrochloric acid) 250mM, KCl (potassium chloride) 375 mM MgCl2 15mM), 2 µl de DTT (dithiothreitol) (0.1M) and wáter, all the mix was incubated at at 37° for two minutes and 1 µl of MMLV(Moloney Murine Leukemia Virus Reverse Transcriptase) Reverse transcriptase- enzyme (200u) (INVITROGEN, Carlsbad, CA) and incubated at 37°C for 50 minutes.

Real-time polymerase chain reaction (qRT-PCR) analysis The mRNA expression levels of the ABCB1 (Hs01069047), and glyceraldehyde 3-phosphate dehydrogenase (GAPDH; Hs00985689) genes were measured using the TaqMan® gene expression assay (Applied Biosystems, Foster City, CA, USA). The GAPDH gene was used as an endogenous control, and each sample was analyzed in triplicate. The relative expression levels were calculated using the 2-ΔΔCtmethod with bone marrow as a calibrator. The high and low expression cut-off points were determined by the mean values observed in healthy donors.

Treatment protocol All the patients recieve an induction remission treatment with an initial pre-induction phase with steroids (prednisone) from day -7 to day -1 (-7 ,-6 = 25mg , -5 , -4 : 50mg , -3, -2: 75mg and on day -1 : 100mg). The induction remission treatment is based on a 28 day treatment with prednisone (60mg/m2),Vincristine (1.5mg/m2 maxium 2mg) and Daunorubicin 60mg/m2 on days +1, +8 and +15. If the patient archive a Complete Remission, continues with a consolidation therapy with sequential blocks of treatment that includes Cytarabine, Etoposide, Methotrexate. If the patient still on remission at the end of consolidation therapy continues on maintenance phase that includes 6-mercaptopurine and a weekly dose of methotrexate for around two years

Response At day 28 of the induction remission treatment, according the result of bone marrow sample the patientes will be declared on remission (less than 5% blast) or refractory (>5% blast cell). If the patient present at any point of treatment an increase on bone marrow blast count the patient is considered on relapse.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* de novo B-cell precursor Acute Lymphoblastic Leukemia
* candidates to first line treatment protocol
* ECOG (Eastern Cooperative Oncology Group) Scale of Performance Status 1/2
* Informed Consent Form for genetic analysis samples
* Precursor B Cell Acute Lymphoblastic Leukemia

Exclusion Criteria:

* Diagnose of Acute Myelogenous Leukemia or Biphenotype Leukemia
* Diagnose of type 2 Diabetes Mellitus
* Previous use of Metformin
* Relapsed Acute Leukemia that require treatment protocol to be started
* Intolerance to prednisone
* ECOG Scale of Performance Status 3/4
* T-cell Acute Lymphoblastic Leukemia
* Philadelphia positive Acute Lymphoblastic Leukemia
* Tumor lysis syndrome at diagnose
* Renal Failure (creatinine leve higher than 2mg/dl)
* Several liver damage (>2 levels de upper normal limit of Aspartate transaminase (AST) and alanine transaminase (ALT)
* Metabolic Acidosis or Lactic Acidosis at diagnose
* Central nervous system infiltration at diagnose
* Extramedullary disease (skin, pleura,eye)
* Active GI bleeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Effect of Metformin on first line treatment Refractoriness in high risk failure ALL patients | 28 day induction remission treatment
  Effect on the refractoriness frequency in high risk failure patients (High levels of ABCB1)
Effect of Metformin on relapse rate and survival of high risk failure ALL patients | 12 months of follow up
  Effect of Metformin on Relapse Free Survival (RFS) on patients with high risk failure (high levels of ABCB1 gene )

REFERENCES:
- [Background] Kim HG, Hien TT, Han EH, Hwang YP, Choi JH, Kang KW, Kwon KI, Kim BH, Kim SK, Song GY, Jeong TC, Jeong HG. Metformin inhibits P-glycoprotein expression via the NF-kappaB pathway and CRE transcriptional activity through AMPK activation. Br J Pharmacol. 2011 Mar;162(5):1096-108. doi: 10.1111/j.1476-5381.2010.01101.x. PMID 21054339
- [Background] Olarte Carrillo I, Ramos Penafiel C, Miranda Peralta E, Rozen Fuller E, Kassack Ipina JJ, Centeno Cruz F, Garrido Guerrero E, Collazo Jaloma J, Nacho Vargas K, Martinez Tovar A. Clinical significance of the ABCB1 and ABCG2 gene expression levels in acute lymphoblastic leukemia. Hematology. 2017 Jun;22(5):286-291. doi: 10.1080/10245332.2016.1265780. Epub 2016 Dec 14. PMID 27960630
- [Derived] Ramos-Penafiel C, Olarte-Carrillo I, Ceron-Maldonado R, Rozen-Fuller E, Kassack-Ipina JJ, Melendez-Mier G, Collazo-Jaloma J, Martinez-Tovar A. Effect of metformin on the survival of patients with ALL who express high levels of the ABCB1 drug resistance gene. J Transl Med. 2018 Sep 3;16(1):245. doi: 10.1186/s12967-018-1620-6. PMID 30176891